CLINICAL TRIAL: NCT01552876
Title: Comparative Clinical Evaluation of Soft Toric Lens Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-4582
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A / nelfilcon A / Filcon II 3 (Other): etafilcon A worn first then nelfilcon A worn second with Filcon II 3 worn third.
  Interventions: Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- nelfilcon A / etafilcon A / Filcon II 3 (Other): nelfilcon A worn first then etafilcon A worn second with Filcon II 3 worn third.
  Interventions: Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3

INTERVENTIONS:
Device: etafilcon A — A daily wear contact lens
  Other Names: 1-DAY ACUVUE MOIST for Astigmatism
Device: nelfilcon A — A daily wear contact lens
  Other Names: Focus Dailies Toric All Day Comfort
Device: Filcon II 3 — a daily disposable
  Other Names: Clariti(TM) 1 day Toric

SUMMARY:
This study is evaluating the initial fit of toric contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be greater than or equal to 18 years old.
* Read, understand, and sign written Statement of Informed Consent.
* Appear able and willing to adhere to the instructions set forth in this clinical protocol.
* Be existing soft contact lens wearers (no extended wear in the last 3 months, but silicone hydrogels in daily wear are allowed).
* Require a visual correction in both eyes (monovision allowed but no monofit).
* Have a spherical contact lens requirement in the range -0.50D to -6.00D.
* Have astigmatism of between -0.50 and -2.00DC in both eyes.
* Monocular distance visual acuity correctable to 6/9 (0.2 logMAR) or better in each eye with best sphero-cylindrical refraction.
* Have normal eyes with no evidence of any ocular abnormality or disease. For the purposes of this study a normal eye is defined as one having: Clear cornea, No anterior segment disorder, No clinically significant slit lamp findings (i.e. oedema, staining, scarring, vascularisation, infiltrates or abnormal opacities), No other active ocular disease or recent surgery

Exclusion Criteria:

* Having worn RGP contact lenses within the last 30 days or PMMA contact lenses within the last 3 months.
* Clinically significant corneal oedema, corneal vascularisation, corneal staining, tarsal abnormalities, bulbar injection or any other abnormality of the cornea that would contraindicate contact lens wear.
* Extended lens wear in last 3 months.
* Any systemic or topical medications that will in the investigator's opinion affect ocular physiology or contact lens performance.
* Any systemic disease affecting ocular health.
* Abnormal lacrimal secretions.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial.
* Any previous anterior ocular surgery.
* Subjects who are known to have an infectious systemic disease (e.g., hepatitis, tuberculosis).
* Subjects who are known to have an immunosuppressive disease (e.g., HIV positive).
* Subjects who are known to have diabetes.
* Employees or family members of the Research site, Principal Investigator or study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Farnham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are considered to be enrolled and not randomized at baseline. There were 42 subjects enrolled and 2 that were not randomized for a study baseline population of 40.
Groups:
- Etafilcon A/ Nelfilcon A/Filcon II 3: etafilcon A worn first, nelfilcon A worn second, Filcon II 3 worn third. Only etafilcon A and nelfilcon A were used in phase I of the study per study protocol, with Filcon II 3 being added to the rotation in Phase II (see outcome 5).
- Nelfilcon A/ Etafilcon A/ Filcon II 3: nelfilcon A worn first, etafilcon A worn second, Filcon II 3 worn third. Only etafilcon A and nelfilcon A were used in phase I of the study per study protocol, with Filcon II 3 being added to the rotation in Phase II (see outcome 5).
Period: Overall Study
Arm/Group | Etafilcon A/ Nelfilcon A/Filcon II 3 | Nelfilcon A/ Etafilcon A/ Filcon II 3
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- All Subjects: All subjects who were enrolled at baseline.
Arm/Group | All Subjects
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.45 (12.707)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Absolute Lens Rotation
Description: At 1-min after lens insertion, lens orientation position was assessed on a scale of 0-180 degree on both eyes.
Time Frame: At 1-min after lens insertion during Phase I
Population: Subjects included in the analysis were those who were enrolled, randomized, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Units Other Than Participants: eyes
Groups:
- Etafilcon A: Those subjects who wore etafilcon A.
- Nelfilcon A: Those subjects who wore nelfilcon A.
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 80 | 80
Degrees | 6.73 [5.29 to 8.56] | 11.38 [8.95 to 14.48]

2. Secondary Outcome: Phase I: Time to Lens Settling
Description: With random insertion and natural blinking, the slit lamp video was used to measure the time of lens settling.
Time Frame: 5 minutes after lens insertion during Phase I
Population: Subjects analyzed were those who were enrolled, randomized, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- Etafilcon A: Those who wore etafilcon A.
- Nelfilcon A: Those who wore nelfilcon A.
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 40 | 40
minutes | 1.60 [1.25 to 2.04] | 1.82 [1.43 to 2.32]

3. Secondary Outcome: Phase I: Number of Blinks Until Settled
Description: Number of blinks for the right eye was counted until lens settling using headcam video.
Time Frame: Baseline to 5 minutes during Phase I
Population: Subjects analyzed are those who were enrolled, randomized, and completed the study.
Measure: Least Squares Mean (Standard Error); unit: Blinks
Arm/Group | Etafilcon A | Nelfilcon A.
Number analyzed (Participants) | 40 | 40
Blinks | 57.29 (6.65) | 74.73 (4.56)

4. Primary Outcome: Phase I: Absolute Lens Rotation
Description: Lens orientation position as assessed on a scale of 0-180 on both eyes.
Time Frame: 3 min after lens insertion during Phase I
Population: Analysis was on those subjects who were enrolled, randomized, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Nelfilcon A
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 80 | 80
Degrees | 6.26 [4.92 to 7.97] | 11.06 [8.70 to 14.07]

5. Other Pre Specified Outcome: Phase II: Absolute Rotation
Description: Absolute rotation of the lens (degrees) at 1-minute post-fit on both eyes. Filcon II 3 lens was only used for comparison in phase II of the study per study protocol.
Time Frame: 1-minute during Phase II
Population: Analysis was on those subjects who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: eyes
Groups:
- Filcon II 3: All subjects wore the Filcon II 3 lens after the wearing of the etafilcon and nelfilcon lenses.
Arm/Group | Etafilcon A | Nelfilcon A | Filcon II 3
Number analyzed (Participants) | 40 | 40 | 40
Number analyzed (eyes) | 80 | 80 | 80
Degrees | 9.99 (14.194) | 17.54 (17.431) | 16.59 (30.820)

ADVERSE EVENTS:
Description: two phases, noted as phase I and phase II
Groups:
- Etafilcon A: Those subjects who wore etafilcon A. (Phase I & II)
- Nelfilcon A: Those subjects who wore nelfilcon A. (Phase I & II)
- Filcon II 3: Those who wore Filcon II 3 during Phase II
Arm/Group | Etafilcon A | Nelfilcon A | Filcon II 3
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days